CLINICAL TRIAL: NCT00677989
Title: The Role of Oxidized Proteins and Free Radicals on Laparoscopic Operation for Perforated Appendicitis
Brief Title: Study on Laparoscopic Operation for Perforated Appendicitis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Heng-Fu Lin, chief of the tramatology division, surgical department, Traumatology Department,Far-Eastern Memorial Hospital, Taipei , Taiwan
Other Study IDs: FEMH No. 96044
Record Dates: First submitted 2008-05-13; First posted 2008-05-15 (Estimated); Last update posted 2009-02-09 (Estimated); Status verified 2009-01

CONDITIONS: Perforated Appendicitis
Keywords: perforated appendicitis; laparoscopic appendectomy; open appendectomy; cytokines; free radicals; oxidized proteins
MeSH Terms: conditions — Appendicitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- LA: LA group: patients with perforated appendicitis treated by laparoscopic operation intentionally
  Interventions: Procedure: Laparoscopic appendectomy
- OA: OA group:patients with perforated appendicitis treated by open approach
  Interventions: Procedure: Open appendectomy

INTERVENTIONS:
Procedure: Laparoscopic appendectomy — laparoscopic appendectomy:did appendectomy by laparoscopic manipulation
  Groups: LA
Procedure: Open appendectomy — open appendectomy: did appendectomy by laparotomy
  Groups: OA

SUMMARY:
The purpose of this study is to conduct a prospective observational study for the open approach and laparoscopic approach for perforated appendicitis. It is also designed to investigate if carbon dioxide pneumoperitoneum will have unwanted effect when treating perforated appendicitis with laparoscopic operation.

DETAILED DESCRIPTION:
The role of laparoscopic appendectomy (LA) for perforated appendicitis is under investigation. According to the results of a previous retrospective study conducted in Far-Eastern Memorial Hospital comparing the clinical outcomes between perforated appendicitis patients treated by laparoscopic and open approach showed favored clinical outcomes for LA. Same as a few studies indicated that laparoscopic appendectomy is a safe and effective procedure for treating patients with perforated appendicitis in terms of hospital stay and wound complications. One the other hand, some authors still concern about the adverse effects of laparoscopy for ruptured appendicitis patients in terms of longer operation time and increased rates of postoperative abscess formation. We hypothesize that prolonged CO2 pneumoperitoneum will produce transient mesenteric ischemic and reperfusion injury when CO2 disinflation, and the free radicals and oxidative proteins provoked by reperfusion injury are responsible for the adverse reaction of LA. The objective of this prospective non-randomized controlled study is to examine the safety and efficacy of laparoscopic appendectomy and compare its outcome with that of the conventional approach for perforated appendicitis patients, with special emphasis on postoperative complication and oxidative stress resulted from pneumoperitoneum..

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted at the emergency station of our hospital expressing pain other than the right lower abdominal quadrant.
* The results of a clinical examination favored the diagnosis of perforated acute appendicitis, and the result of abdominal computed tomography revealed signs of acute appendicitis and intra-abdominal fluid accumulation.
* Patients were accepted to our study only if perforated appendicitis remained as the most likely diagnosis of their condition and if they were between 12 from 80 years old with informed consent.

Exclusion Criteria:

* Age less than 12 years
* older than 80 years
* perforated appendicitis was not revealed by pathologic investigation
* diverticulitis being diagnosed during surgery
* pelvic inflammatory disease or other gynecologic disease found during laparoscopic examination or diagnosed before operation
* the patient declining to enroll in this study

Ages: 12 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with perforated appendicitis treated at the Far-Eastern Memorial Hospital, Taipei,Taiwan
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2008-05; Primary Completion 2010-12 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
paraoperative outcomes | till patients are discharged

SECONDARY OUTCOMES:
levels of paraoperative serum cytokines, free radicals, and oxidized proteins. | since preoperative preparation till 48 hours after operation

CONTACTS AND LOCATIONS:
Overall Officials: Heng-Fu Lin, MD, Principal Investigator — Traumatology division, Surgical department, Far-Eastern Memorial Hospital
Locations (1):
- Surgical Department, Far-Eastern Memorial Hospital, Taipei, Taiwan

REFERENCES:
- [Background] Semm K. Endoscopic appendectomy. Endoscopy. 1983 Mar;15(2):59-64. doi: 10.1055/s-2007-1021466. PMID 6221925
- [Background] Chung RS, Rowland DY, Li P, Diaz J. A meta-analysis of randomized controlled trials of laparoscopic versus conventional appendectomy. Am J Surg. 1999 Mar;177(3):250-6. doi: 10.1016/s0002-9610(99)00017-3. PMID 10219865
- [Background] Garbutt JM, Soper NJ, Shannon WD, Botero A, Littenberg B. Meta-analysis of randomized controlled trials comparing laparoscopic and open appendectomy. Surg Laparosc Endosc. 1999 Jan;9(1):17-26. PMID 9950122
- [Background] Golub R, Siddiqui F, Pohl D. Laparoscopic versus open appendectomy: a metaanalysis. J Am Coll Surg. 1998 May;186(5):545-53. doi: 10.1016/s1072-7515(98)00080-5. PMID 9583695
- [Background] Sauerland S, Lefering R, Holthausen U, Neugebauer EA. Laparoscopic vs conventional appendectomy--a meta-analysis of randomised controlled trials. Langenbecks Arch Surg. 1998 Aug;383(3-4):289-95. doi: 10.1007/s004230050135. PMID 9776459
- [Background] Temple LK, Litwin DE, McLeod RS. A meta-analysis of laparoscopic versus open appendectomy in patients suspected of having acute appendicitis. Can J Surg. 1999 Oct;42(5):377-83. PMID 10526524
- [Background] Frazee RC, Bohannon WT. Laparoscopic appendectomy for complicated appendicitis. Arch Surg. 1996 May;131(5):509-11; discussion 511-3. doi: 10.1001/archsurg.1996.01430170055010. PMID 8624197
- [Background] Klingler A, Henle KP, Beller S, Rechner J, Zerz A, Wetscher GJ, Szinicz G. Laparoscopic appendectomy does not change the incidence of postoperative infectious complications. Am J Surg. 1998 Mar;175(3):232-5. doi: 10.1016/s0002-9610(97)00286-9. PMID 9560127
- [Background] So JB, Chiong EC, Chiong E, Cheah WK, Lomanto D, Goh P, Kum CK. Laparoscopic appendectomy for perforated appendicitis. World J Surg. 2002 Dec;26(12):1485-8. doi: 10.1007/s00268-002-6457-7. Epub 2002 Sep 26. PMID 12297916
- [Background] Lin HF, Wu JM, Tseng LM, Chen KH, Huang SH, Lai IR. Laparoscopic versus open appendectomy for perforated appendicitis. J Gastrointest Surg. 2006 Jun;10(6):906-10. doi: 10.1016/j.gassur.2005.12.012. PMID 16769550
- [Background] Martin LC, Puente I, Sosa JL, Bassin A, Breslaw R, McKenney MG, Ginzburg E, Sleeman D. Open versus laparoscopic appendectomy. A prospective randomized comparison. Ann Surg. 1995 Sep;222(3):256-61; discussion 261-2. doi: 10.1097/00000658-199509000-00004. PMID 7677456
- [Background] Yao CC, Lin CS, Yang CC. Laparoscopic appendectomy for ruptured appendicitis. Surg Laparosc Endosc Percutan Tech. 1999 Aug;9(4):271-3. PMID 10871175
- [Background] Joris J, Cigarini I, Legrand M, Jacquet N, De Groote D, Franchimont P, Lamy M. Metabolic and respiratory changes after cholecystectomy performed via laparotomy or laparoscopy. Br J Anaesth. 1992 Oct;69(4):341-5. doi: 10.1093/bja/69.4.341. PMID 1419439
- [Background] Cho JM, LaPorta AJ, Clark JR, Schofield MJ, Hammond SL, Mallory PL 2nd. Response of serum cytokines in patients undergoing laparoscopic cholecystectomy. Surg Endosc. 1994 Dec;8(12):1380-3; discussion 1383-4. doi: 10.1007/BF00187340. PMID 7878501